CLINICAL TRIAL: NCT06953102
Title: The Prevalence and Association of Anxiety and Sleep Disturbances Among Medical Students: A Cross-sectional Study
Brief Title: Prevalence and Association of Anxiety and Sleep Disturbances Among Medical Students.
Status: Completed | Type: Observational
Sponsor: Government Medical College, Patiala (Other Government)
Responsible Party: Principal Investigator, Yuvraj Kaushal, Dr. Yuvraj Kaushal, Government Medical College, Patiala
Other Study IDs: Trg.9(310)2024/13198-201
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disturbances; Anxiety
Keywords: Sleep disturbances.; Anxiety; Medical students; Pittsburgh Sleep Quality Index (PSQI); Beck Anxiety Inventory (BAI); Sleep quality
MeSH Terms: conditions — Parasomnias; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phase-2 MBBS Students: The group included in Phase-2 MBBS Students i.e. 2nd year students in med school
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — Survey was conducted to collect their responses to PSQI and BAI questionnaires.

SUMMARY:
Observational, Cross-sectional study

DETAILED DESCRIPTION:
It was a cross-sectional study conducted in December 2024 with the consent of 200 undergraduate medical students of a tertiary care hospital affiliated medical college, who qualified as per the inclusion criteria.

Inclusion criteria:

All the students of MBBS Phase-II.

Exclusion criteria:

Students with prior diagnosed Sleep disorders Students with prior diagnosed co-morbidities Students unable/unwilling to answer the question.

ELIGIBILITY:
Inclusion criteria:

- All the students of MBBS Phase-II.

Exclusion criteria:

* Students with prior diagnosed Sleep disorders
* Students with prior diagnosed co-morbidities
* Students unable/unwilling to answer the question.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students of MBBS
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Sleep Disturbances | 1 month
  The Pittsburgh Sleep Quality Index (PSQI) has been used to assess the pattern and the quality of sleep.[8] This questionnaire assesses sleep quality over a 1-month time interval based on self-report by the participant. PSQI differentiates 'Poor' from 'Good' sleep by measuring Seven Domains: Subjective Sleep Quality, Latency, Sleep Duration, Sleep Efficiency, Disturbances, Medication, and Daytime Dysfunction over the last month. The measure consists of 19 individual items, creating 7 components that produce one global score and take 5-10 minutes to complete.
Assessment of Anxiety | 1 month
  To assess Anxiety, the Beck Anxiety Inventory (BAI)[9] has been used. This scale is a self-report measure of anxiety in children and adults, which asks the subject to rate 21 items on a scale of 0-3. The questions used in this measure ask the subject about common symptoms of anxiety that the subject had had during the past week. It is designed for individuals aged 17 and above and takes 5-10 minutes to complete. The total score is calculated by the standard mean of the responses to the 21 items. A score of 0-21 = low anxiety. A score of 22-35 = moderate anxiety. A Score of 36 and above signifies potentially concerning levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuvraj Kaushal, Patiāla, Punjab, India

IPD SHARING:
Plan to Share IPD: No
Participant Confidentiality

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT06953102/SAP_000.pdf